

# "Comparative Study of Clinical Outcomes and Safety between Colistin and Tigecycline for Multi-Drug Resistant Gram Negative Bacteria."

## **Protocol study**

Submitted for fulfillment Philosophy of Doctoral Degree in Pharmaceutical sciences (Clinical Pharmacy)

# **Submitted by:**

#### Nada Abd El-Hamed Saad

Clinical Pharmacist
Under supervision of

## Dr. Raghda Roshdy Sayed Hussein

Assistant Professor and Acting Head of Department of Clinical Pharmacy Faculty of Pharmacy, Beni-Suef University

## Dr. Shaymaa Nafady Abdelfattah

Lecturer of Gastroenterology, Hepatology and Infectious diseases Faculty of Medicine, Beni-Suef University

# **Dr. Yasmin Mohamed Madany**

Lecturer of Clinical Pharmacy Faculty of Pharmacy, Beni-Suef University

#### Dr. Marwa Mohsen Mahmoud

Lecturer of Clinical Pharmacy Faculty of Pharmacy, Beni-Suef University

> Faculty of Pharmacy Beni-suef University 2024

# Comparative Study of Clinical Outcomes and Safety between Colistin and Tigecycline for Multi-Drug Resistant Gram Negative Bacteria.

#### I. Introduction:

The Centers for Disease Control and Prevention (CDC) and the European Center for Disease Prevention and Control have defined Multi-drug resistant (MDR) Gram-negative bacteria as acquired non-susceptibility to at least one drug in three or more antimicrobial categories. Extensively drug-resistant (XDR) Gram-negative bacteria was defined as non-susceptibility to at least one agent in all but two or fewer antimicrobial categories (i.e. bacterial isolates remain susceptible to only one or two categories). Pan drug-resistant (PDR) was defined as non-susceptibility to all agents in all antimicrobial categories (1).

MDR, XDR and PDR of Escherichia coli, Klebsiella pneumoniae, Enterobacter spp., Acinetobacterbaumannii, and Pseudomonas aeruginosa have been known by difficult-to-treat (DTT) infections that not respond to treat with as  $\beta$ -lactams, including carbapenems, extended-spectrum cephalosporins such as ceftazidime, ceftriaxone, and cefepime and  $\beta$ -lactam/  $\beta$ -lactamase inhibitor combinations, and fluoroquinolones(2).

In the past few decades, bacteria developed various mechanisms of resistance to almost available antibiotics as tetracycline, beta-lactams, fluoroquinolones and aminoglycosides. Colistin and tigecycline have become the last treatment for MDR gram negative bacteria(3)(2).

Colisin is polymyxin E antibiotic. Colistin has a unique mechanism of action against MDR and XDR bacteria regardless of the resistance. Colistin has an antimicrobial activity against aerobic Gram-negative bacteria(4). Colistin is the last choice treatment for life-threatening infections, such as carbapenem-resistant P. aeruginosa, E. coli, A. baumannii, K. pneumoniae, and other Enterobacteriaceae(3).

Although, colistin has a good antimicrobial activity against MDR and XDR, some old literatures reported that colistin associated with high side effects as neuorotoxicity, neuromuscular blockade, hematoxicity and nephrotoxicity and mortality risk (5)(6). In 1970, the use of colistin was limited for treatment patients with cystic fibrosis only. Latterly, some new studies reported that colistin's side

effects are less common than old studies and they resolved after discontinuation of colistin in severe cases (7).

Tigecycline belongs to a tetracycline class that used for the treatment of MDR infections (gram negative and gram positive bacteria). In 2005, the Food and Drugs Administration (FDA) approved tigecycline that administrated in a parenteral form. The FDA reported in 2010 that the treatment with tigecycline was associated with high risk for mortality (8). Recently, tigecycline has been used for treatment complicated intra-abdominal infections (CIAI), complicated skin and skin structures infections (CSSTI) with the exclusion of diabetes foot infection, and community-acquired bacterial pneumonia (CAP) as monotherapy in adult(9).

The FARES and the clinical trial studies suggested that tigecycline administration associated with gastrointestinal symptoms (nausea, vomiting and diarrhea), pancreatitis, increased hepatic function, jaundice, cholestatic, bleeding risk, thrombocytopenia and Steven-Johnson syndrome(8)(10).

The objective of this study to prospectively compare between the clinical outcomes and safety of colistin and tigecycline in patients with MDR gram negative bacteria in Intensive Care Unit.

# II. Aim and objectives:

Objective from this study to compare the clinical outcomes and safety between colistin and tigecycline for multi-drug resistant gram negative bacteria.

#### III. Method and material:

## **Study site:**

Study will be in Beni-Suef university hospital.

# **Study design:**

Prospective randomized controlled study. The method of randomization was a sealed envelope technique.

## **Study duration:**

The study will be conducted from December 2024 to May 2025.

### **Study population:**

- **Group I**: 66 patients received intravenous **colistin** 300 mg colistin base activity (CBA) as **loading dose**, **followed by** 2.5–5mg/kg/day of CBA in 2 divided doses as **a maintenance dose** in intensive care unit to treat their MDR infection.(11)
- **Group II**: 66 patients received intravenous **tigecycline**100 mg single dose as **loading dose**, followed by 25-50 mg every 12 hours **maintenance dose** in intensive care unit to treat their MDR infection(12).

### Sample size technique:

Sample size was calculated using G\*Power (3.1.9.4) software for windows using Fisher analysis test. A total sample size of 132 participants was estimated for 95% power, α- error probability 0.05. Analysis of data was performed using IBM SPSS v. 25 (Statistical Package for Social science) for Windows.

### **Sample size calculation:**

**Exact** - Proportions: Inequality, two independent groups (Fisher's exact test)

**Options:** Exact distribution

Analysis: A priori: Compute required sample size

**Input:** Tail(s) = Two

Proportion p1 = 0.58Proportion p2 = 0.261  $\alpha$  err prob = 0.05Power (1- $\beta$  err prob) = 0.95Allocation ratio N2/N1 = 1

**Output:** Sample size group 1 = 66

Sample size group 2 = 66 Total sample size = 132

Actual power = 0.9501125Actual  $\alpha$  = 0.0316077

### **Inclusion criteria:**

Study will include adult patient (male, female), (age from 18 to 70 years) admitted to intensive care unit in study period (six months) who received intravenous colistin or tigecycline as antimicrobial drug for treatment their MDR gram negative infection (13).

## **Exclusion criteria:**

- Patient admitted to intensive care unit younger than 18 years or older than 70 years (14).
- Liver transplantation patients.
- Patients are chronic kidney disease (CKD on hemodialysis or baseline creatinine clearance (crcl) < 10 ml/min (estimated by Cockcroft Gault equation).
- Patients received renal replacement therapy before or during admission.
- Patient is on any other nephrotoxic drug (vancomycin, aminoglycosides, NSAIDs, cyclosporine, amphotericin B, etc.) (Aggarwal & Dewan, 2018).
- Pregnant and lactating women (16).
- Patients refused the consent of the study.

# **Study procedure:**

- Demographic and medical history for all patients included in this study will be recorded.
- Complete physical examination for all patients included in this study will be taken.
- Basic routine investigation for all patients included in this study will be measured as Complete blood Count test (CBC), blood pressure and temperature.
- Improvement of signs and symptoms after the end of antibiotic course as temperature.
- **Renal function** tests will be measured **before** patients received colistin or tigecycline and **after 72 hours from first dose**:

- > Serum creatinine level (scr).
- **Hepatic function** tests will be measured **before** patients received colistin or tigecycline and **after 72 hours from first dose:** 
  - ➤ Alanine transaminase (ALT)
  - ➤ Aspartate transaminase (AST)
  - > Serum total bilirubin (TBIL)
- 14 days Survival rate after starting colistin or tigecycline will be recorded.
- The severity of the illness will be assessed by using the Acute Physiology and Chronic Health Evaluation II (APACHE II) scoring system will be calculated.(Wu et al., 2022).

#### **Statistical analysis:**

All statistical analysis will be performed by using SPSS version 23. The demographic and clinical characteristics of patients will be expressed as mean  $\pm$  standard deviation (SD). Student's t-tests or Mann-Whitney tests will be used to compare between groups. Chi-square tests or exact tests (Fisher's exact test or likelihood ratio test) will be used to detect the existence of association between variables.

## **Ethical consideration:**

An ethical approval will be obtained from ethical committee of Faculty of medicine Beni-Suef University.

All patients in study agree to participate of their own free will and that they have been fully informed regarding the procedures of the research project and any potential risks.

If any patient included in study want to withdraw, stop study in this patient immediately.

The study will start after approval of the research ethical committee and according to guideline of the Declaration of Helsinki.

#### **IV.** References:

- 1. Kadri SS, Adjemian J, Lai YL, Spaulding AB, Ricotta E, Rebecca Prevots D, et al. Difficult-to-treat resistance in gram-negative bacteremia at 173 US hospitals: Retrospective cohort analysis of prevalence, predictors, and outcome of resistance to all first-line agents. Clinical Infectious Diseases. 2018;67(12):1803–14.
- 2. Abushanab D, Nasr ZG, Al-Badriyeh D. Efficacy and Safety of Colistin versus Tigecycline for Multi-Drug-Resistant and Extensively Drug-Resistant Gram-Negative Pathogens—A Meta-Analysis. Antibiotics. 2022 Nov 1;11(11).
- 3. El-Sayed Ahmed MAEG, Zhong LL, Shen C, Yang Y, Doi Y, Tian GB. Colistin and its role in the Era of antibiotic resistance: an extended review (2000–2019). Vol. 9, Emerging Microbes and Infections. Taylor and Francis Ltd.; 2020. p. 868–85.
- 4. Falagas ME, Kyriakidou M, Voulgaris GL, Vokos F, Politi S, Kechagias KS. Clinical use of intravenous polymyxin B for the treatment of patients with multidrug-resistant Gram-negative bacterial infections: An evaluation of the current evidence. Vol. 24, Journal of Global Antimicrobial Resistance. Elsevier Ltd; 2021. p. 342–59.
- 5. Yahav D, Farbman L, Leibovici L, Paul M. Colistin: New lessons on an old antibiotic. Vol. 18, Clinical Microbiology and Infection. Blackwell Publishing Ltd; 2012. p. 18–29.
- 6. Shatri G, Tadi P. Polymyxin. 2024.
- 7. Andrade FF, Silva D, Rodrigues A, Pina-Vaz C. Colistin update on its mechanism of action and resistance, present and future challenges. Vol. 8, Microorganisms. MDPI AG; 2020. p. 1–12.
- 8. Kaewpoowat Q, Ostrosky-Zeichner L. Tigecycline: A critical safety review. Vol. 14, Expert Opinion on Drug Safety. Informa Healthcare; 2015. p. 335–42.
- 9. Yaghoubi S, Zekiy AO, Krutova M, Gholami M, Kouhsari E, Sholeh M, et al. Tigecycline antibacterial activity, clinical effectiveness, and mechanisms and epidemiology of resistance: narrative review. Available from: https://doi.org/10.1007/s10096-020-04121-1
- 10. Huang YT, Yu CI, Chen PY, Wang CC, Wu CC. Comparison of bleeding risk between colistin—tigecycline and colistin—carbapenem treatment regimens: A retrospective cohort study. Infect Drug Resist. 2021;14:4949–55.
- 11. Lee YJ, Wi YM, Kwon YJ, Kim SR, Chang SH, Cho S. Association between Colistin Dose and Development of Nephrotoxicity. Crit Care Med. 2015 Jun 20;43(6):1187–93.
- 12. Yaghoubi S, Zekiy AO, Krutova M, Gholami M, Kouhsari E, Sholeh M, et al. Tigecycline antibacterial activity, clinical effectiveness, and mechanisms and epidemiology of resistance: narrative review. Available from: https://doi.org/10.1007/s10096-020-04121-1
- 13. Wu S, Wu G, Wang X, Jiang H, Wu H. A study of clinical characteristics and risk factors of mortality associated with tigecycline. 2022; Available from: https://doi.org/10.21203/rs.3.rs-1603424/v1

- 14. Cheng A, Chuang YC, Sun HY, Sheng WH, Yang CJ, Liao CH, et al. Excess Mortality Associated with Colistin-Tigecycline Compared with Colistin-Carbapenem Combination Therapy for Extensively Drug-Resistant Acinetobacter baumannii Bacteremia: A Multicenter Prospective Observational Study. Crit Care Med. 2015 Jun 20;43(6):1194–204.
- 15. Aggarwal R, Dewan A. Comparison of nephrotoxicity of Colistin with Polymyxin B administered in currently recommended doses: A prospective study. Ann Clin Microbiol Antimicrob. 2018 Mar 23;17(1).
- 16. Fan G, Jin L, Bai H, Jiang K, Xie J, Dong Y. Safety and Efficacy of Tigecycline in Intensive Care Unit Patients Based on Therapeutic Drug Monitoring [Internet]. 2020. Available from: http://journals.lww.com/drug-monitoring